CLINICAL TRIAL: NCT03747913
Title: Effect of Oxidative Stress on Acute Exercise-induced Mobilization and Apoptosis of Hematopoietic, Endothelial and Mesenchymal Stem and Progenitor Cells and Mature Endothelial Cells in Healthy Young Male Subjects
Brief Title: Oxidative Stress as an Acute Exercise-induced Mechanism of Stem and Progenitor Cell Mobilization
Acronym: EISMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EISMO
Record Dates: First submitted 2018-11-12; First posted 2018-11-20 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Each participant enrolled in the study will be part of the supplementation and control condition group in a non-randomized order
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antioxidative Supplementation (Experimental): Each participant conducts two identical cycling tests, first without and a week later with antioxidative supplementation
  Interventions: Dietary Supplement: Antioxidative supplementation

INTERVENTIONS:
Dietary Supplement: Antioxidative supplementation — Each participant conducts two identical cycling tests, first without and a week later with antioxidative supplementation

SUMMARY:
It is already known from literature that exercise mobilizes stem and progenitor cells into the peripheral blood. However, the exact mechanisms thereof remain to be fully elucidated.

The investigators hypothesize that exercise-induced oxidative stress could be at least one of the responsible mechanisms and therefore want to study the exercise-induced stem and progenitor cell mobilization in a group of healthy young men when they exercise with, compared to when they exercise without antioxidative supplementation.

The primary outcome is numbers of stem and progenitor cells in the peripheral blood after an acute bout of exercise. As a secondary outcome, numbers of apoptotic mature and immature cells in the blood will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* Healthy
* Normal Body-Mass-Index (BMI): 18.5-24.9 kg∙m-2
* Active (fulfill World Health Organization-guidelines for recommended levels of physical activity for adults aged 18 - 64 years)
* Willing to adhere to the study rules

Exclusion Criteria:

* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders etc. of the participant
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Regular intake of medication
* Regular intake of antioxidant supplementations

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in exercise-dependently mobilized stem and progenitor cell numbers in the peripheral blood with antioxidative supplementation | On visit 2 after the exercise test without supplementation and then again on visit 3 after the exercise test with prior supplementation (1 week)
  Numbers of hematopoietic, endothelial and mesenchymal stem and progenitor cells and mature endothelial cells in the peripheral blood will be measured after an acute bout of exercise first without and then with prior antioxidative supplementation.

SECONDARY OUTCOMES:
Changes in numbers of exercise-induced apoptotic cells and oxidative stress markers in the peripheral blood with antioxidative supplementation | On visit 2 after the exercise test without supplementation and then again on visit 3 after the exercise test with prior supplementation (1 week)
  Numbers of apoptotic mononuclear cells, apoptotic hematopoietic, endothelial and mesenchymal stem and progenitor cells and apoptotic mature endothelial cells, as well as in oxidative stress markers in the peripheral blood will be measured after an acute bout of exercise first without and then with prior antioxidative supplementation.

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Physiology Lab, Institute of Human Movement Sciences and Sport, ETH Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Schmid M, Martins HC, Schratt G, Kropfl JM, Spengler CM. MiRNA126 - RGS16 - CXCL12 Cascade as a Potential Mechanism of Acute Exercise-Induced Precursor Cell Mobilization. Front Physiol. 2021 Dec 9;12:780666. doi: 10.3389/fphys.2021.780666. eCollection 2021. PMID 34955891